CLINICAL TRIAL: NCT02370381
Title: Vergleich Zwischen Hb Und INR Aus Nsaenblut Und venösem Blut
Brief Title: Hemoglobin and INR Out of Nose Blood
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SM_16_02_2015
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nose blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epistaxis: Patients with active anterior epistaxis

SUMMARY:
Nose bleeding (epistaxis) is a common emergency. It is often difficult to estimate blood loss and the current hemoglobin of patients. In patients with oral anticoagulation, it is important to measure the level of hemodilution. Several situations with the importance of the fast determination of these parameters have been identified in previous studies [1,2]. The blood sampling from the venous punction is the standard in these investigations. However, this requires the corresponding painful puncture and also the time required at the laboratory.

Since many patients present themselves with active bleeding, it is obvious that this blood could be used for determining the following parameters: Hemoglobin and INR/Quick. The nose blood can be analyzed with commercial rapid test devices. If these devices could generate same or similar results and after further validation of the method, painful punctures could be waived.

DETAILED DESCRIPTION:
Patients with active epistaxis are verbally elucidated about the study and the verbal consent is obtained. According to the agreement a few drops of nose blood are preserved. Subsequently the standard therapy is performed. This blood sample is promptly analyzed with the rapid test devices.

We successfully applied the exception to the analysis of blood samples prior to obtaining the written consent due to following reasons: Analysis with the rapid test devices needs to be immediate and without delay in order to satisfy quality standards prescribed by the manufacturers. In addition, patient's treatment should not be delayed.

Simultaneously, a venous blood sample for the corresponding values is carried out according to medical indications. After the treatment of the acute emergency and thus after the greatest stress situation, we ask the patient again whether he agrees to the study conditions. The written consent is obtained in the end of the acute treatment.

Both inception and termination of the research project will be reported within 90 days of the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active nose bleeding
* Indication for routine blood sampling
* Aged 18 to 99 years
* Verbal informed consent before implementation takes place
* Written consent of the participating person after investigation and completion of treatment

Exclusion Criteria:

* No active bleeding
* Routine blood sampling for medical reasons not indicated
* Lack of understanding of the study or investigation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential candidates with active epistaxis are recruited consecutively at the Polyclinic.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin in gram/liter and INR/Quick in % | During the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soyka, Dr. med., Principal Investigator — ORL USZ
Locations (1):
- Zurich University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Soyka MB, Holzmann D. Should we test the prothrombin time in anticoagulated epistaxis patients? Allergy Rhinol (Providence). 2013 Spring;4(1):e52-3. doi: 10.2500/ar.2013.4.0049. PMID 23772329
- [Background] Murer K, Ahmad N, Roth BA, Holzmann D, Soyka MB. THREAT helps to identify epistaxis patients requiring blood transfusions. J Otolaryngol Head Neck Surg. 2013 Jan 31;42(1):4. doi: 10.1186/1916-0216-42-4. PMID 23663751